CLINICAL TRIAL: NCT07199127
Title: Novel Endoscopic Classification for Duodenal Polyposis in Individuals With Familial Adenomatous Polyposis
Brief Title: Duodenal Polyposis Classification in FAP
Acronym: DRACO
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: IRCCS Ospedale San Raffaele (Other)
Responsible Party: Sponsor
Other Study IDs: IRB# INT-12/18
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Duodenum Cancer; Familial Adenomatous Polyposis; Duodenal Polyposis; Ampulla of Vater Adenoma; FAP Gene Mutation; FAP; Duodenal Neoplasms; Duodenal Adenoma; Ampulla of Vater Cancer
Keywords: Spigelman; Duodenal Polyposis
MeSH Terms: conditions — Duodenal Neoplasms; Adenomatous Polyposis Coli

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Individuals with duodenal advanced neoplasia (Training cohort): Individuals who developed biopsy-confirmed duodenal or ampullary high-grade dysplasia (HGD) or adenocarcinoma after the index EGD, within the training cohort (aka, cases)
  Interventions: Diagnostic Test: DRACO
- Individuals with duodenal advanced neoplasia (validation cohort): Individuals who developed biopsy-confirmed duodenal or ampullary high-grade dysplasia (HGD) or adenocarcinoma after the index EGD, within the validation cohort (aka, cases)
  Interventions: Diagnostic Test: DRACO
- Individuals with duodenal advanced neoplasia (Testing cohort): Individuals who developed biopsy-confirmed duodenal or ampullary high-grade dysplasia (HGD) or adenocarcinoma after the index EGD, within the testing cohort (aka, cases)
  Interventions: Diagnostic Test: DRACO
- Individuals without duodenal advanced neoplasia (Training cohort): Individuals who remained free from duodenal or ampullary high-grade dysplasia and adenocarcinoma after the index EGD, within the training cohort (aka, controls)
  Interventions: Diagnostic Test: DRACO
- Individuals without duodenal advanced neoplasia (Validation cohort): Individuals who remained free from duodenal or ampullary high-grade dysplasia and adenocarcinoma after the index EGD, within the validation cohort (aka, controls)
  Interventions: Diagnostic Test: DRACO
- Individuals without duodenal advanced neoplasia (Testing cohort): Individuals who remained free from duodenal or ampullary high-grade dysplasia and adenocarcinoma after the index EGD, within the testing cohort (aka, controls)
  Interventions: Diagnostic Test: DRACO

INTERVENTIONS:
Diagnostic Test: DRACO — A novel endoscopic classification to predict the risk of duodenal and ampullary high-grade dysplasia and cancer from baseline esophagogastroduodenoscopy (EGD)
  Other Names: Duodenal Risk Assessment in adenomatous polyposis Coli Oncogene

SUMMARY:
Duodenal cancer is the leading cause of cancer-related mortality in patients with familial adenomatous polyposis (FAP), yet the current Spigelman staging system provides limited predictive accuracy for advanced neoplasia. The DRACO study (Duodenal Risk Assessment in adenomatous polyposis Coli -Oncogene) is a multicenter, STROBE- and CONSORT-compliant cohort study that analyzes upper endoscopies from genetically confirmed FAP patients across independent cohorts to develop, validate, and externally test two multivariable risk models.

DETAILED DESCRIPTION:
Duodenal cancers represent the leading cause of cancer-related mortality in individuals with familial adenomatous polyposis (FAP). While endoscopic surveillance is a critical component of duodenal cancer management, clinical decisions are primarily guided by the Spigelman staging system. Introduced in 1989, this framework stratifies patients into four stages based on duodenal polyp size, number, histology, and the grade of dysplasia.

Despite its widespread use, the Spigelman system was not originally designed to predict cancer incidence or progression and lacks formal validation for these outcomes. A recent systematic review and meta-analysis confirmed its limited sensitivity for detecting duodenal cancers, at approximately 50%, with even lower sensitivity for papillary cancer. This limitation in early cancer detection also constrains the identification of patients at elevated risk of malignant transformation during a window in which endoscopic intervention might still be feasible. As high-grade dysplasia (HGD) is a well-established precursor to adenocarcinoma and a valid therapeutic target, the inability of the current system to anticipate HGD and its progression to cancer can undermine opportunities for timely, minimally invasive intervention.

The current clinical paradigm reserves prophylactic surgery or intensified endoscopic therapy primarily for patients with Spigelman stage IV disease. However, both cancer and high-grade dysplasia frequently arise in patients with lower-stage disease. Given the already limited sensitivity of the Spigelman system for cancer detection, its sensitivity for predicting the development of HGD is likely even lower. Consequently, relying on a stage IV threshold may delay preventive intervention beyond the window of opportunity for feasible endoscopic management.

These limitations have led to a growing recognition of the need to revise the Spigelman classification system. Two broad strategies have been proposed to improve its clinical utility: reweighting the existing components to better reflect their prognostic contribution, or integrating patient-level variables, such as age and desmoid tumor status, to more accurately capture individual risk trajectories. Importantly, a staging system intended to guide endoscopic surveillance should prioritize prevention by informing timely intervention before malignant transformation occurs. Therefore, risk stratification must be grounded in the likelihood of developing pre-cancerous lesions, such as high-grade dysplasia, not solely on the risk of overt carcinoma. The DRACO study was designed to fill this gap in knowledge.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed germline diagnosis of FAP, as defined by genetic testing
* Two or more upper gastrointestinal endoscopies
* Complete documentation of all Spigelman classification variables at each endoscopic evaluation

Exclusion Criteria:

* Histological grading of duodenal polyps incomplete
* Follow-up data were unavailable
* Duodenal surgery before study baseline endoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with familial adenomatous polyposis, defined by a pathogenic/likely pathogenic germline Adenonomatous Polyposis Coli (APC) gene variant, undergoing surveillance for duodenal polyposis using esophagogastroduondeoscopy (EGD)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-02-02 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2030-01-15 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | Through study completion, on average 5 years
  True Positivity Rate: the probability of a positive test result, conditioned on the individual truly developing duodenal or ampullary high-grade dysplasia or adenocarcinoma

SECONDARY OUTCOMES:
Specificity | Through study completion, on average 5 years
  True Negative Rate: the probability of a negative test result, conditioned on the individual being truly free from duodenal or ampullary high-grade dysplasia or adenocarcinoma
Proportion of correct predictions (true positives and true negatives) among the total cases (i.e., accuracy) | Through study completion, on average 5 years
  A measure of trueness: proportion of correct predictions (both true positives and true negatives) among the total number of cases examined

CONTACTS AND LOCATIONS:
Overall Officials: Marco Vitellaro, M.D., Study Chair — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (2):
- Italy (2):
  - IRCCS Ospedale San Raffaele, Milan, MI
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan

IPD SHARING:
Plan to Share IPD: Undecided
Data collected for the study will be made available to others, including de-identified participant data, at publication, via a signed data access agreement and at the discretion of the investigators' upon approval of the proposed use of such data

REFERENCES:
- [Background] Bulow S, Christensen IJ, Hojen H, Bjork J, Elmberg M, Jarvinen H, Lepisto A, Nieuwenhuis M, Vasen H. Duodenal surveillance improves the prognosis after duodenal cancer in familial adenomatous polyposis. Colorectal Dis. 2012 Aug;14(8):947-52. doi: 10.1111/j.1463-1318.2011.02844.x. PMID 21973191
- [Background] Zaffaroni G, Mannucci A, Koskenvuo L, de Lacy B, Maffioli A, Bisseling T, Half E, Cavestro GM, Valle L, Ryan N, Aretz S, Brown K, Buttitta F, Carneiro F, Claber O, Blanco-Colino R, Collard M, Crosbie E, Cunha M, Doulias T, Fleming C, Heinrich H, Huneburg R, Metras J, Nagtegaal I, Negoi I, Nielsen M, Pellino G, Ricciardiello L, Sagir A, Sanchez-Guillen L, Seppala TT, Siersema P, Striebeck B, Sampson JR, Latchford A, Parc Y, Burn J, Moslein G. Updated European guidelines for clinical management of familial adenomatous polyposis (FAP), MUTYH-associated polyposis (MAP), gastric adenocarcinoma, proximal polyposis of the stomach (GAPPS) and other rare adenomatous polyposis syndromes: a joint EHTG-ESCP revision. Br J Surg. 2024 May 3;111(5):znae070. doi: 10.1093/bjs/znae070. PMID 38722804
- [Background] Mannucci A, Puzzono M, Goel A, Moslein G, Balafas S, Di Serio MS, Cavestro GM. The Spigelman Staging System and the Risk of Duodenal and Papillary Cancer in Familial Adenomatous Polyposis: A Systematic Review and Meta-Analysis. Am J Gastroenterol. 2024 Apr 1;119(4):617-624. doi: 10.14309/ajg.0000000000002688. Epub 2024 Jan 31. PMID 38294150
- [Result] Karstensen JG, Bulow S, Hojen H, Jelsig AM, Jespersen N, Andersen KK, Wewer MD, Burisch J, Pommergaard HC. Cancer in Patients With Familial Adenomatous Polyposis: A Nationwide Danish Cohort Study With Matched Controls. Gastroenterology. 2023 Sep;165(3):573-581.e3. doi: 10.1053/j.gastro.2023.05.010. Epub 2023 May 16. PMID 37201686